CLINICAL TRIAL: NCT05932134
Title: The Effects of High Protein Supplementation, Core Muscle Rehabilitation and Neuromuscular Electrostimulation (NMES) Programs on Clinical Outcomes in Patients With Prolonged Mechanical Ventilation (PMV〕
Brief Title: High Protein, Core Muscle Rehab, Muscular Electrostimulation in Prolonged Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202300154A3
Record Dates: First submitted 2023-04-26; First posted 2023-07-06 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2024-08

CONDITIONS: Prolonged Mechanical Ventilation; Protein Deficiency
MeSH Terms: conditions — Protein Deficiency | interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: Participants will randomly stratify into four groups: (1) Usual care (UC), (2) UC + high protein diet (HP), (3) UC + HP + core muscle rehabilitation, (4) UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES).
  Researchers will compare group 2,3,4 to control group (1, usual care) to see if high protein diet, core muscle rehabilitation, neuromuscular electric stimulation works.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Usual care (No Intervention): Usual care as RCC protocol in Chang Gung Memorial hospital
- UC + high protein diet (HP) (Experimental): The HP groups will maintain unchanged total daily caloric intake and increasing protein content to 1.5g/kg/day.
  Interventions: Dietary Supplement: UC + high protein diet (HP)
- UC + HP + core muscle rehabilitation (Experimental): Protein provision was not reduced in case of renal failure. Core muscle rehabilitation is sitting on bedside with or without aids, for 30 minutes, twice per day, 5 days per week, for 3 weeks.
  Interventions: Behavioral: UC + HP + core muscle rehabilitation
- UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES) (Experimental): NMES was applied for 30 min, twice per day, 5 days per week, for 3 weeks via surface rectangular electrodes. Electrodes were placed on back designed to activate latissimus dorsi and abdominal wall designed to activate the transversus abdominis and internal and external oblique muscles. Electrical muscle stimulation was performed by using a commercial stimulator (GEMORE, GM300E, Taipei, Taiwan) with biphasic waves at a simulation frequency of 30 Hz and pulse width of 400s, cycling 2s on and 4s off. Electrical muscle stimulation intensity was gradually increased until a visible muscle contraction was observed (median 60 mA [range 50-65 mA].
  Interventions: Device: UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES)

INTERVENTIONS:
Dietary Supplement: UC + high protein diet (HP) — The HP groups will maintain unchanged total daily caloric intake and increasing protein content to 1.5g/kg/day.
  Arms: UC + high protein diet (HP)
Behavioral: UC + HP + core muscle rehabilitation — Core muscle rehabilitation is sitting on bedside with or without aids, for 30 minutes, twice per day, 5 days per week, for 3 weeks
  Arms: UC + HP + core muscle rehabilitation
Device: UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES) — NMES was applied for 30 min, twice per day, 5 days per week, for 3 weeks via surface rectangular electrodes. Electrodes were placed on back designed to activate latissimus dorsi and abdominal wall designed to activate the transversus abdominis and internal and external oblique muscles. Electrical muscle stimulation was performed by using a commercial stimulator (GEMORE, GM300E, Taipei, Taiwan) with biphasic waves at a simulation frequency of 30 Hz and pulse width of 400s, cycling 2s on and 4s off. Electrical muscle stimulation intensity was gradually increased until a visible muscle contraction was observed (median 60 mA [range 50-65 mA].
  Arms: UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES)

SUMMARY:
The goal of this clinical trial is to learn about in patients with prolong mechanical ventilation. This main questions aims to answer are:

* High protein formula intake benefit in successful weaning from ventilator
* Core muscle rehabilitation benefit in successful weaning from ventilator
* neuromuscular electric stimulation benefit in successful weaning from ventilator

Participants will receive high protein diet, core muscle rehabilitation, neuromuscular electric stimulation (NMES).

Researchers will compare patients with interventions to control group to see if high protein diet, core muscle rehabilitation, neuromuscular electric stimulation works.

DETAILED DESCRIPTION:
The investigator aims to investigate the efficacy of below list methods in patients with prolong mechanical ventilator:

* High protein formula intake benefit in successful weaning from ventilator
* Core muscle rehabilitation benefit in successful weaning from ventilator
* neuromuscular electric stimulation benefit in successful weaning from ventilator

Participants will randomly stratify into four groups: (1) Usual care (UC), (2) UC + high protein diet (HP), (3) UC + HP + core muscle rehabilitation, (4) UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES).

Researchers will compare group 2,3,4 to control group (1, usual care) to see if high protein diet, core muscle rehabilitation, neuromuscular electric stimulation works.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 20 year old
2. using mechanical ventilator for more than 21 days (including patients under tracheostomy or endotracheal tube)
3. stable clinical condition, without using inotropic agent (arterial blood gas pH : 7.35-7.45, PaO2≥60 mm Hg at FiO2 40%, absence of signs and symptoms of uncontrolled infection, and hemodynamic stability)
4. maximal inspiratory pressure (MIP) < 30mmHg
5. under enteral nutrition (EN) via NG tube.

Exclusion Criteria:

1. Acute infection and sepsis (fever up to 38.5 degree)
2. Severe neuromuscular disease, or uncontrolled epilepsy
3. Bony fracture or DVT history
4. Wound over the abdomen
5. Congestive heart failure with EF < 40% or using pacemaker
6. BMI>35 kg/M2, or severe edema
7. Patients with hepatic failure, rapid progressed malignancy, or pregnancy were also excluded.
8. Under parenteral nutrition (PN)
9. Use pacemaker

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Yu Lin, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang SW, Lin HC, Chou YF, Lin TY, Lo CY, Huang HY, Fang YF, Hsieh MH, Lin SM, Lo YL, Hsieh MJ, Kao KC, Lin CY, Huang CC. The Impact of Higher Protein Intake in Patients with Prolonged Mechanical Ventilation. Nutrients. 2022 Oct 20;14(20):4395. doi: 10.3390/nu14204395. PMID 36297079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The inclusion criteria were as follows: 1. age ≥ 20 year old, 2. latest 21 days after their admission into the ICU, using mechanical ventilator for more than 21 days , 3. stable clinical condition, 4. maximal inspiratory pressure (MIP) < 30mmHg, 5. under enteral nutrition (EN) via NG tube.
  We obtained written informed consent from the patients or their legally acceptable surrogate.
Pre-assignment Details: According to the order of enrollment, patients will be randomly assigned into four groups: (1) Usual care (UC) + high protein diet (HP), (2) UC + HP + core muscle rehabilitation, (3) UC + HP + core muscle rehabilitation + neuromuscular electrostimulation (NMES) (4) UC. Patients were randomized accordingly using a table of random numbers and sealed envelopes. After randomization, on the first three day, we initiated interventions and maintained intervention for 21 days.
Period: Overall Study
Arm/Group | Usual Care | UC + High Protein Diet (HP) | UC + HP + Core Muscle Rehabilitation | UC + HP + Core Muscle Rehabilitation + Neuromuscular Electric Stimulation (NMES)
Started | 10 | 30 | 30 | 30
Completed | 8 | 26 | 28 | 29
Not Completed | 2 | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total 100 patients were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | UC + High Protein Diet (HP) | UC + HP + Core Muscle Rehabilitation | UC + HP + Core Muscle Rehabilitation + Neuromuscular Electric Stimulation (NMES) | Total
Number analyzed (Participants) | 10 | 30 | 30 | 30 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We had analyze the difference of age between groups.
  years | 72.8 (10.9) | 69.3 (11.9) | 67.2 (12.1) | 71.5 (9.1) | 69.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We had analyze the sex ratio between groups.
  Participants
    Female | 2 | 14 | 14 | 11 | 41
    Male | 8 | 16 | 16 | 19 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
modified Nutrition Risk in Critically ill (NUTRIC) score [Mean (Standard Deviation); unit: units on a scale] — a scoring system for nutrition status evaluation in critical illness patients. (including age, APACHE II, SOFA, comorbidities, Days from hospital to ICU admission) 5-0 =>High Score (Associated with worse clinical outcomes (mortality, ventilation), These patients are the most likely to benefit from aggressive nutrition therapy.) 0-4 =>LOW Score (These patients have a low malnutrition risk) Population: We analyze the mNUTRIC score (range 0-10) between groups.
  units on a scale | 5.3 (1.3) | 5.1 (1.4) | 4.8 (1.8) | 5.4 (1.8) | 5.1 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Weaning Rate
Description: weaning success defined as weaning from ventilator for 5 consecutive days
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual care | UC + high protein diet (HP) | UC + HP + core muscle rehabilitation | UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES)
Number analyzed (Participants) | 10 | 30 | 30 | 30
Participants | 3 | 20 | 22 | 26

2. Secondary Outcome: In Hospital Mortality
Description: through the end of admission, up to 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual care | UC + high protein diet (HP) | UC + HP + core muscle rehabilitation | UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES)
Number analyzed (Participants) | 10 | 30 | 30 | 30
Participants | 3 | 5 | 5 | 4

3. Secondary Outcome: Length of Mechanical Ventilator Usage
Description: total ventilator use days in this admission
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual care | UC + high protein diet (HP) | UC + HP + core muscle rehabilitation | UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES)
Number analyzed (Participants) | 10 | 30 | 30 | 30
days | 74.4 (27.1) | 56.5 (24.1) | 57.1 (29.9) | 41.1 (12.9)

4. Secondary Outcome: Length of ICU Stay
Description: total ICU stay in this admission
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual care | UC + high protein diet (HP) | UC + HP + core muscle rehabilitation | UC + HP + core muscle rehabilitation + neuromuscular electric stimulation (NMES)
Number analyzed (Participants) | 10 | 30 | 30 | 30
days | 31.3 (12.8) | 25.7 (7.9) | 26.0 (8.3) | 23.7 (7.5)

ADVERSE EVENTS:
Time Frame: from enrollment through the end of the admission, up to 3 months
Description: adverse event defined as related to the intervention. If the mortality was not happened during intervention period or directly related to the intervention, it's not defined as adverse events of this study.
Arm/Group | Usual Care | UC + High Protein Diet (HP) | UC + HP + Core Muscle Rehabilitation | UC + HP + Core Muscle Rehabilitation + Neuromuscular Electric Stimulation (NMES)
All-Cause Mortality (participants affected / at risk) | 3/10 | 5/30 | 5/30 | 4/30
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
First, our trial is a single-center trial made in RCC. The nutritional protocol, interventions were not blinded to the staff, which may possibly introduce bias. Moreover, we calculated caloric intake and protein intake using body weight as ESPEN guideline. We didn't use calorimetry to predict precisely energy consumption. The nutrition need might be not adequate for patients. This study enrolled relatively small number of subjects in each group, which may limit the validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT05932134/Prot_SAP_000.pdf